CLINICAL TRIAL: NCT00164554
Title: Fetal Alcohol Syndrome/ARND Research Consortion-Oklahoma
Brief Title: Fetal Alcohol Syndrome/ARND Research Consortion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Oklahoma (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CDC-NCBDDD-3813; U84/CCU020163-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2008-04-28 (Estimated); Status verified 2005-09

CONDITIONS: Fetal Alcohol Syndrome
Keywords: treatment; control
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

INTERVENTIONS:
Behavioral: Parent-child Interaction Therapy (PCIT)

SUMMARY:
Children will receive comprehensive evaluations through the UOHSC ABC program The assessment for the child will include: medical issues (including medication), dysmorphic examination, intellectual assessment, academic achievement, language, and motor skills. This program will provide appropriate non-study services and referrals. Eligible families will be randomly assigned to treatment group or control group. Treatment group will receive Parent Child Interaction Therapy (PCIT). The Control group will receive standard referrals and services through the ABC program and the parent education/advocacy component of the project.

DETAILED DESCRIPTION:
PCIT has been adapted by the applicant for group administration. The intervention will consist of 90-minute sessions of PCIT once a week for 14 weeks. During PCIT sessions parents and children will participate in activities that promote interactions. A behavior specialist who will be observing through a two-way mirror assists parents in development of appropriate behaviors and interaction techniques. Parents will be prompted by use of in-ear devices (i.e., bug in the ear). This intervention has been shown to be effective in other populations. For each family, individualized goals for parent-child interactions will be set and reviewed each session. Homework assignments also will be given.

Parent Component: Three 90-minute sessions conducted in a group format. Topics will include: FAS/ARND education, impact of FAS/ARND on families, specific development of a child with FAS/ARND, and FAS/ARND social skills and deficits.

Evaluation Plan: Treatment and control groups will be compared using pre- and post-tests measures. Post-tests will be at the conclusion of the intervention and at a 6, 12, and 18-month follow-ups. Process (e.g., parent satisfaction, compliance, etc) and outcome (e.g., behavior, family functioning, etc) measures will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3 to 7 years

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100
Dates: Start 2001-10; Study Completion 2005-06

PRIMARY OUTCOMES:
compliance with directives

CONTACTS AND LOCATIONS:
Overall Officials: John Mulvihill, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States